CLINICAL TRIAL: NCT03479086
Title: Defining the Clinical Role of Topiramate in the Treatment of Alcohol Dependence in Australia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South West Sydney Local Health District (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Professor Paul Haber, Principle Clinical Investigator, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X16-0231
Record Dates: First submitted 2018-03-05; First posted 2018-03-27 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Topiramate; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topiramate (Experimental): Topiramate 200mg/day
  Interventions: Drug: Topiramate
- Naltrexone (Experimental): Naltrexone 50mg/day
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Topiramate — 200mg/day 100mg b.i.d
  Arms: Topiramate
Drug: Naltrexone — 50mg/day
  Arms: Naltrexone

SUMMARY:
To compare the clinical effectiveness, tolerability, and cost-effectiveness of topiramate to active control (naltrexone) on treatment outcomes for alcohol dependence in a double-blind randomised controlled trial.

DETAILED DESCRIPTION:
Clinicians urgently require new treatment strategies for the treatment of alcohol dependence. Although alcohol use disorders are a leading cause of preventable death in Australia, their treatment is generally not evidence based. The medications currently approved for use in Australia for the management of alcohol dependence have limited efficacy, and existing research does not address the heterogeneity of treatment response.

Targeted personalised medicine addresses this heterogeneity with better medicine selection for patients based on their genotype and clinical comorbidities.

Members of our research team have recently demonstrated findings that support the use of topiramate (TOP) 200 mg/day to reduce heavy drinking and pharmacogenetic findings that implicate the GluK1 receptor subunit in the mechanism of these effects.

This project will evaluate the clinical effectiveness and tolerability of topiramate relative to the active control naltrexone (NTX) in heavy drinkers.

Investigators hypothesise that topiramate treated patients will be better able to achieve a reduction in heavy drinking and predict that, based on prior research, that the effects would be moderated by a single nucleotide polymorphism (rs2832407) in GRIK1.

Research personnel will utilise an innovative prospective pharmacogenetic randomisation approach to a double-blind, randomised, controlled trial.

Individuals will receive 12 weeks of titrated treatment with topiramate (200 mg/day) or naltrexone (50mg/day) and medical management.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Use Disorder according to the Diagnostic and Statistical Manual of Mental Disorders Version V criteria
* Age 18-70
* Average weekly alcohol consumption of >30 standard drinks for men and >25 standard drinks for women, with a weekly average of > 2 heavy drinking days during the month before screening
* Adequate cognition and English language skills to give valid consent and complete research interviews
* Willingness to give written informed consent
* Willingness to provide a blood sample for genotyping
* Written informed consent

Exclusion Criteria:

* Active major psychological disorder associated with psychosis, significant suicide risk, and signs of impaired cognitive functioning
* Pregnancy or lactation
* Concurrent use of any psychotropic medication other than antidepressants
* Currently taking any tricyclic antidepressant
* Use of antiretroviral dolutegravir
* Any substance dependence other than nicotine
* Opioid abuse, opioid dependence, or on opioid maintenance treatment
* Clinically significant liver disease
* History of nephrolithiasis
* History of glaucoma
* Lack of stable housing and/or contact phone number
* Previous hypersensitivity to TOP or NTX
* Any alcohol pharmacotherapy within the past month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of heavy drinking days, as measured by the Time Line Follow Back | Over 12 weeks
  Corroborated with Phosphatidylethanol (PEth) levels
Time to relapse, as measured by the Time Line Follow Back | Over 12 weeks
  Corroborated with PEth levels
Time to lapse, as measured by the Time Line Follow Back | Over 12 weeks
  Corroborated with PEth levels
Number of days abstinent, as measured by the Time Line Follow Back | Over 12 weeks
  Corroborated with PEth levels
Number of standard drinks per drinking day, as measured by the Time Line Follow Back | 12 weeks
  Corroborated with PEth levels

SECONDARY OUTCOMES:
Self report of adverse events | 12 weeks
  as reported by patient during weekly medical management sessions facilitated by the treating doctor.
Penn Alcohol Craving Scale for alcohol craving | 12 weeks
  as measured by amount of time spent thinking and craving for alcohol, difficulty in resisting consumption of alcohol if present and hypothetical pleasure associated with consumption of alcohol.
DASS21 score for presence and/or severity of anxiety | 12 weeks
  as measured by cumulative score of anxiety related questions on the Depression, Anxiety Stress Scale-21 (DASS21).
DASS21 score for presence and/or severity of depression | 12 weeks
  as measured by cumulative score for depression related questions
Insomnia Severity Index for sleep disturbances | 12 weeks
  as measured by cumulative score of satisfaction with current sleep patterns and extent to which sleep disturbances interfere and impair with every day activities and daily functioning
Blood glucose test for diabetes | 12 weeks
  as measured by fasting blood glucose levels in blood
Liver function tests for clinical markers of liver injury | 12 weeks
  as measured by levels of liver enzymes, Alanine Transaminase (ALT), Alkaline Phosphatase (ALP) and Aspartate Transaminase (AST) in blood
Body Mass Index | 12 weeks
  as measured by weight in kilograms (kg) and height in metres (m). These two measurements will be combined together to report BMI in kg/m^2.
Number of cigarettes smoked daily, as measured by Time Line Follow Back | 12 weeks
Self report of daily measures of expectancies, confidence and drinking | 12 weeks
  as measured using a scale of the likelihood of having a good time and feeling more relaxed if alcohol was consumed.

OTHER OUTCOMES:
The moderating effect of the OPRM1 polymorphism in response to naltrexone, as measured by number of heavy drinking days | 12 weeks
Cost-effectiveness of topiramate versus naltrexone, as measured by Disability-Adjusted Life Years (DALYs) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Haber, MBBS, Principal Investigator — Sydney Local Health District; Andrew Baillie, PhD, Principal Investigator — Macquarie University; Kirsten C Morley, PhD, Principal Investigator — University of Sydney
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Logge WB, Haber PS, Hurzeler T, Gallagher H, Kranzler H, Morley KC. Neural cue reactivity and intrinsic functional connectivity in individuals with alcohol use disorder following treatment with topiramate or naltrexone. Psychopharmacology (Berl). 2025 Jul;242(7):1641-1652. doi: 10.1007/s00213-025-06745-7. Epub 2025 Jan 24. PMID 39853353
- [Derived] Morley KC, Kranzler HR, Luquin N, Baillie A, Shanahan M, Trent R, Teesson M, Haber PS. Topiramate versus naltrexone for alcohol use disorder: study protocol for a genotype-stratified, double-blind randomised controlled trial (TOP study). Trials. 2018 Aug 16;19(1):443. doi: 10.1186/s13063-018-2824-z. PMID 30115121